CLINICAL TRIAL: NCT04626024
Title: Safety And Efficacy Of Tyrosine Kinase Inhibitor Cessation For Chronic Myeloid Leukemia Patients With Stable Molecular Response In A Real World Population
Brief Title: Safety And Efficacy Of TKI Cessation For CML Patients With Stable Molecular Response In A Real World Population
Acronym: TOKIN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Martha Mims, Professor of Medicine; Section Chief, Hematology/Oncology, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-48054
Record Dates: First submitted 2020-10-16; First posted 2020-11-12 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Chronic Myeloid Leukemia; Chronic Myeloid Leukemia, BCR/ABL-Positive, in Remission; Chronic Myeloid Leukemia in Remission
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate; Dasatinib; nilotinib; bosutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- All Subjects Enrolled (stop taking TKI) (Experimental): Patients with a diagnosis of Philadelphia chromosome- or BCR-ABL1-positive CML (as determined by cytogenetics, FISH, or PCR), prior evidence of a quantifiable BCR-ABL1 transcript by RT-PCR, and whom have been taking TKI for > 36 months with a current status of complete molecular remission (CMR). TKI cessation begins within 7 days of study registration. Patients undergo BCR-ABL1 test every month in 24 months.
  Interventions: Other: Imatinib Mesylate, Dasatinib, Nilotinib or Bosutinib Withdrawal; Drug: Imatinib Mesylate, Dasatinib, Nilotinib or Bosutinib Re-initiation

INTERVENTIONS:
Other: Imatinib Mesylate, Dasatinib, Nilotinib or Bosutinib Withdrawal — Stop taking TKI medication
Drug: Imatinib Mesylate, Dasatinib, Nilotinib or Bosutinib Re-initiation — Re-start TKI medication
  Other Names: Gleevec; Sprycel; Tasigna; Bosulif

SUMMARY:
This is a single-arm, phase II study to evaluate safety and efficacy of tyrosine kinase inhibitor (TKI) cessation for chronic myeloid leukemia (CML) patients with stable molecular response in a real world population.

DETAILED DESCRIPTION:
Transitioning from busulfan, hydroxyurea, IFN-α to tyrosine kinase inhibitors (TKIs) has dramatically altered the natural history of CML. Patients with CML appropriately managed with TKIs are able to benefit from near normal life expectancy. Given the age-adjusted incidence of 1.6 per 100,000 people combined with a reduced annual mortality of less than 2% to 3% per year, it is expected the prevalence in the US to increase from approximately 70,000 in 2010 to a projected 144,000 in 2030. Thus, advancing our knowledge regarding clinical management is critical in order to care for this expanding population.

However the morbidity associated with prolonged TKI exposure remains a substantial burden on this patient population. In addition to a relatively benign side effect profile (edema, muscle cramps, diarrhea, nausea, musculoskeletal pain, rash and other skin problems, abdominal pain, fatigue, joint pain, and headaches), patients continued to experience grade 3 and 4 adverse events (neutropenia, thrombocytopenia, anemia, elevated liver enzymes, congestive heart failure, and other drug-related adverse events) more than 2 years after initiating therapy. For patients with high-risk CML that may benefit from faster and/or deeper molecular responses, or who develop intolerance or resistance to imatinib, second generation TKIs (dasatinib, nilotinib, and bosutinib) are available. Indeed, there is a structural and dose-dependent relationship between TKIs and ischemic heart disease, ischemic cerebrovascular events and/or peripheral artery disease accompanied with a linear increase in the cumulative frequency of these cardiovascular events over time. Additionally, experts believe the cost of CML medicines "are too high, are unsustainable, may compromise access of needy patients to highly effective therapy, and are harmful to the sustainability of our national health care systems." Given the implications on quality of life, adverse events and financial burden on patients, TKI therapy should be discontinued when medically appropriate.

Thankfully, discontinuation of TKIs in CML-CP patients with RT-PCR negative for BCR-ABL1 transcripts (Undetectable Minimal Residual Disease, UMRD) or MR has established that 38% to 45% of patients are able to achieve TFR with persistence of UMRD and MR at 5 and 8 years, respectively. Subsequent studies (EURO-SKI, ENESTfreedom, ENESTop, and DADI) have independently validated these results, and patients who experience MR will mostly do so within three to six months after discontinuation.

Furthermore, in patients with complete cytogenetic response, those who have a deeper molecular response (>3 log reduction in transcripts) compared to those without have an improved estimated 7-year event-free survival. ddPCR is a powerful tool that allows for the absolute quantitation of nucleic acids and provides a more precise and sensitive assay than real-time PCR (RT-PCR) in detecting BCR-ABL1 transcripts. There is neither a precise molecular mechanism to characterize MR, nor a clinically actionable assay to determine which patients will benefit from TKI cessation and achieve TFR. Thus, leveraging ddPCR can impact patient outcomes in CML-CP patients undergoing TKI treatment by potentially determining who is expected to achieve of TFR.

Cancer causing mutations can affect oncogenes that normally stimulate growth, suppressor genes that normally inhibit growth, and repair genes that normally limit mutations. Of the 20,000 protein coding genes in the human genome, approximately ~140 genes can promote tumorigenesis while the remaining passenger mutations confer no selective growth advantage. In CML, genomic analysis has identified variants in patients with poor outcomes. Therefore, mutational analysis of clinically relevant genes and genes of emerging clinical relevance could provide insight into which patients are at risk for relapse.

Prior to these findings, a truly curable clinical status after CML diagnosis was previously attainable only with allogeneic stem cell transplantation. It is known that successful remission in relapsing CML patients who have undergone stem cell transplantation was primarily driven by an alloreactive T-cell dependent graft-versus-leukemia effect. The cytotoxic role of a WT-1 peptide specific TCR Vβ21 T-cell clone against K562 cells has been demonstrated in vitro. Taken together, these data suggest a role of immune cells and the subsequent maturation, generation, and homing of CML-antigen-specific T-lymphocytes - the hallmark of elimination during cancer immune surveillance. Massively paralleled sequencing of the complementarity determining region 3 by TCR-sequencing (TCR-seq) allows for a detailed understanding of the T-cell repertoire and is representative of clonal distribution, antigenic response diversity, and the degree of T-cell immunomodulation. A diverse T-cell repertoire capable of recognizing CML-specific antigens with concomitant clonal expansion may be associated with successful TFR and potentially provide additional biomarkers towards identifying patients with CML-CP who should be optimal candidates for TKI cessation.

ELIGIBILITY:
Inclusion Criteria

1. Patients who are 18 years or older
2. Patients have a diagnosis of Philadelphia chromosome- or BCR-ABL1-positive CML (as determined by cytogenetics, FISH, or PCR).
3. Prior evidence of a quantifiable BCR-ABL1 transcript by RT-PCR
4. Patients who have been taking TKI for > 36 months.
5. Patients must have a history of stable molecular response, defined as MR4.5 for ≥24 months, as documented by ≥3 separate tests performed at least three months apart.
6. Patient must have a current status of complete molecular remission (CMR), defined as MR4.5 (per section 5.1), within 30 days of signing consent.
7. ECOG performance status < 2
8. Patients must have normal marrow function within 30 days of registration, as defined:

   * Absolute Neutrophil Count (ANC) ≥ 1.5 x 10E9/L
   * Hemoglobin ≥ 9.0 g/dL
   * Platelets ≥ 100 x 10E9/L
9. Patients must not have any signs of extramedullary leukemia
10. Patients must have a life expectancy of more than 12 months in the absence of any intervention
11. All participants must be informed of the investigational nature of this study and must sign and give written informed consent
12. Contraception requirements will be as per routine clinical practice.

Exclusion Criteria

1. Patients who are unable or unwilling to give their consent to participate to the study.
2. Previous or planned allogeneic stem cell transplantation
3. Patients who have pathologies or treatments that are able to enhance the potential relapse risk after stopping Imatinib.
4. Patient has received an investigational agent within last 2 years
5. Atypical BCR-ABL transcript not quantifiable by standard RQ-PCR.
6. Patient cannot have had a known interruption of TKI therapy of greater than 14 consecutive days or for a total of 6 weeks in the six months prior to registration.
7. Another primary malignant disease, except those that do not currently require treatment (adequately treated conditions, such as excised skin cancer or cervical intra-epithelial neoplasia would not be considered exclusion criteria. If in doubt, please refer to the Principal Investigator).
8. Any medical condition that, in the opinion of the investigator, would exclude the patient from participating in this study.
9. Active liver disease (e.g., chronic active hepatitis, cirrhosis).
10. Known diagnosis of human immunodeficiency virus (HIV) infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-12-22 (Actual); Primary Completion 2028-11-15 (Estimated); Study Completion 2028-11-15 (Estimated)

PRIMARY OUTCOMES:
Molecular relapse (MR) free survival | From date of TKI cessation to the date of MR or censoring, assessed up to 6 months
  The Kaplan-Meier method will be used to estimate MR free survival rate at 6 months after TKI cessation with a 95% confidence interval.

SECONDARY OUTCOMES:
ddPCR of BCR-ABL1 values affecting MR free survival | At baseline (just before TKI cessation begins)
  ddPCR of BCR-ABL1 values (copies/μl) at baseline (just before TKI cessation begins) will be assessed by Cox proportional hazard regression model.
Event free survival (EFS) | From date of TKI cessation to the date of the event defined or censoring, assessed at 6 months and up to 24 months
  The event for EFS is defined as any of the following events: (i) loss of complete hematologic response (CHR), (ii) to accelerated phase or blast crisis (AP/BC), (iii) death due to any cause, whichever occurs first.The Kaplan-Meier method will be used to estimate EFS at 6months and up to 24 months after TKI cessation with a 95% confidence interval.
Progression-free survival (PFS) | From date of TKI cessation to the date of the progression defined or censoring, assessed at 6 months and up to 24 months
  The event of progression is defined by AP/BC or death due to any causes, whichever occurs first. The Kaplan-Meier method will be used to estimate PFS at 6 months and up to 24 months after TKI cessation with a 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Martha P. Mims, MD, PhD, Principal Investigator — Baylor College of Medicine
Locations (4):
- United States (4):
  - Baylor College of Medicine- McNair Campus, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - CHI St. Luke's Health Baylor College of Medicine Medical Center, Houston, Texas
  - Harris Health System- Smith Clinic, Houston, Texas

IPD SHARING:
Plan to Share IPD: No